CLINICAL TRIAL: NCT00536562
Title: Comprehensive Cardiac Rehabilitation Programming For Patients Following Transient Ischemic Attack
Brief Title: Cardiac Rehabilitation for TIA Patients
Acronym: CR-TIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-07-251
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: TIA (Transient Ischemic Attack)
Keywords: Comprehensive Cardiac Rehabilitation; Randomized Controlled Trial; TIA (Transient Ischemic Attack); Mild Non-Disabling Stroke; Vascular Protection
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual Care as provided through the Stroke Prevention Clinic
- Cardiac Rehabilitation (Active Comparator): Usual Care plus Comprehensive Cardiac Rehabilitation Program
  Interventions: Behavioral: Comprehensive Cardiac Rehabilitation (CR)

INTERVENTIONS:
Behavioral: Comprehensive Cardiac Rehabilitation (CR) — 6-month Comprehensive Cardiac Rehabilitation program consisting of: 1) initial medical assessment by case manager and physician to determine CR strategies; 2) entry exercise stress test; 3) multi-disciplinary assessment and intervention to achieve risk factor targets in nutrition & psychological services as needed; 4) twice per week supervised exercise training and twice per week home-based exercise following an individualized, progressive prescription; 5) Exit assessment at 6 months.
  Other Names: Cardiac Rehabilitation
  Arms: Cardiac Rehabilitation

SUMMARY:
The purpose of this study is to determine, in patients following a TIA, whether a 6-month case-managed exercise based multi-factorial cardiac rehabilitation program (CR), similar to those used in patients following a heart attack, can significantly improve exercise capacity, reduce cholesterol, reduce depression, and improve thinking ability.

DETAILED DESCRIPTION:
Similar risk factors predispose patients to both cardiovascular and cerebrovascular events. Two hundred consecutive patients from Stroke Prevention Clinics (SPC) at London Health Sciences Centre and the Ottawa Hospital (100 patients from each site) who have sustained a Transient Ischemic Attack (TIA) or mild non-disabling stroke will participate in a randomized controlled trial in which they will either receive Usual Care (UC) as delivered by the SPC, or enter the existing multi-disciplinary 6-month comprehensive cardiac rehabilitation (CR) intervention at LHSC and Ottawa in addition to receiving UC. This study seeks to determine the benefits of providing a CR program to TIA/mild non-disabling stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented TIA or mild non-disabling stroke within the previous 3 months.
* At least one of the following vascular risk factors: hypertension, ischemic heart disease, diabetes mellitus, dyslipidemia or cigarette smoking

Exclusion Criteria:

* Inability to speak or understand English or provide informed consent.
* Severe aphasia that renders communication difficult or impossible.
* Modified Rankin Scale score of greater than or equal to 3.
* Mini-Mental Status Examination score of less than or equal to 20.
* Evidence of intracranial hemorrhage confirmed by CT scan or MRI study.
* Anticipated or recent (<30 days) carotid endarterectomy, angioplasty and/or stenting.
* Resides >1 hour travel time from London or Ottawa.
* Prior participation in a CCR program.
* Inability to perform expected exercise training of CCR program.
* Evidence of cardioembolic source for TIA/stroke such as atrial fibrillation, valvular disease, septal defect or left ventricular wall motion abnormality.
* Participation in another clinical trial that could interfere with the intervention or outcomes of the current study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-09; Primary Completion 2014-06-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
To determine compared to usual care, whether a 6-month CR strategy results in significant improvements of functional capacity, lipid profile, depression symptoms and cognition. | 6 months

SECONDARY OUTCOMES:
Outcomes include cerebrovascular and cardiovascular events, pre-post changes in physiological, anthropometric and behavioral vascular risk factors, neurocognitive measures, and quality of life. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neville G. Suskin, MBChB, MSc, Principal Investigator — University of Western Ontario & London Health Sciences Centre
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario